CLINICAL TRIAL: NCT01335516
Title: Follow-up of Glypressin (Terlipressin) Clinical Efficacy in the Treatment of Bleeding Oesophageal Varices
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: FE999908 CS04
Record Dates: First submitted 2011-04-07; First posted 2011-04-14 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Gastrointestinal Bleeding; Oesophageal Varices
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Esophageal and Gastric Varices | interventions — Terlipressin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Glypressin (terlipressin) — Study drug (without placebo)

SUMMARY:
Terlipressin is an effective and safe treatment for bleeding caused by rupture of oesophageal varices, which are life-threatening complications of liver cirrhosis.

Oesophageal varices are abnormal dilatation of veins occurring in the lower oesophagus, which can develop in patients with cirrhosis. Bleeding caused by rupture of these varices is a life-threatening complication with mortality between 20-50%.

Such bleeding can be treated with drug therapy and/or endoscopic; endoscopic therapy consists of a flexible tube equipped with a camera at the terminal end, allowing for visualizing and treating the oesophageal varices.

In this study, investigators will evaluate the safety and efficacy of terlipressin - Glypressin 1 mg, powder and solvent for solution for injection.

The non-interventional observational study "Follow-up of Glypressin (terlipressin) clinical efficacy in the treatment of bleeding oesophageal varices" aims to demonstrate that administration of Glypressin (terlipressin 1 mg) controls the bleeding in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients that present an important upper gastrointestinal bleeding, being suspected or diagnosed of liver cirrhosis, with bleeding oesophageal varices visualized endoscopically.

(An important upper gastrointestinal bleeding is one requiring at least 2 units/24h of transfused blood).

Exclusion Criteria:

* Septic shock
* Patients with recent history of coronary insufficiency
* Uncontrolled arterial hypertension
* Chronic respiratory failure
* Symptomatic arteritis
* Chronic renal failure
* Pregnant women
* Hypersensitivity to terlipressin
* Patients with body weight below 55 kg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 estimated eligible participants with an age of 18-70 years, suspected or diagnosed with bleeding oesophageal varices. Patients have cirrhosis (from any cause, any Child class) and upper gastrointestinal haemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical efficacy of Glypressin: measured by rapid control of heamorrhage; reduced mortality post-haemorrhage | Up to 6 months
  Vital signs (blood pressure, heart rate, and body temperature) and routine safety lab analysis
To evaluate the safety profile of Glypressin: measured by number of patients with adverse events | Up to 6 months

SECONDARY OUTCOMES:
To evaluate/monitor the ease of administration in ER | Up to 6 months
  Easiness of use in ER (easy to reconstitute, easy to administer, flexible dosage)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Emergency County Hospital - Surgery Clinic No.1, Târgu Mureş, Mureș County, Romania